CLINICAL TRIAL: NCT03103308
Title: Effects of a Multidirectional Walking Program on Physical Function and Quality of Life in Hematopoetic Stem Cell Transplant Patients
Brief Title: Hematopoetic Stem Cell Transplant and Physical Function
Acronym: HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20160711
Record Dates: First submitted 2017-03-17; First posted 2017-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Cancer; Walking
Keywords: Cancer; Exercise; Physical Function
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walk training and transplant (Experimental): Multidirectional walk training with activity monitoring after bone marrow transplant
  Interventions: Other: Walk Training and Transplant
- Activity Monitoring and transplant (Experimental): Activity monitoring alone after bone marrow transplant.
  Interventions: Other: Activity Monitoring and Transplant

INTERVENTIONS:
Other: Walk Training and Transplant — Subjects will receive free activity monitors and have three training sessions per week for the duration of their bone marrow transplant treatment
  Arms: Walk training and transplant
Other: Activity Monitoring and Transplant — Subjects will receive free activity monitors for the duration of their bone marrow transplant treatment
  Arms: Activity Monitoring and transplant

SUMMARY:
This study will determine if a structured walking intervention will help maintain or improve physical activity levels, physical function and quality of life in hematopoietic stem cell transplant patients.

DETAILED DESCRIPTION:
The researchers will quantify the decline in physical function of HSCT patients using valid and reliable tests aimed to mimic activities of daily living, quantify cardiovascular health, and quantify muscle power declines. Also, patients will undergo a walking program during their hospitalization, which is designed to increase physical activity levels and maintain and improve physical function and quality of life. Additionally, using valid and reliable questionnaires, the researchers will gauge perception of exercise, quantify current exercise levels, determine preference of exercise programs and counseling, and measure differences in quality of life before and after HSCT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be between 40 and 80 years of age
* Willing and able to provide written informed consent in English
* Ability to comprehend the purpose of the study
* Be scheduled to receive an autologous or allogeneic hematopoietic stem cell transplant at Sylvester Comprehensive Cancer Center
* Have an expected hospital stay of at least 2 weeks
* Not currently be participating in an exercise training program

Exclusion Criteria:

* Dementia, altered mental status, or psychiatric condition
* Received erythropoiesis-stimulating proteins within 4 weeks prior to enrollment
* Comorbid conditions that would contraindicate exercise testing
* Undergoing concurrent non-transplant-related chemotherapy or radiation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
The Physical Performance Test Battery | 10 minutes
  Physical Function

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy: Bone Marrow Transplant Questionaire Related Quality of Life | 20 minutes
  Health-related quality of Life
Patient Reported Outcome Measurement Information System | 20 minutes
  Health Related Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Sylvester Comprehensive Cancer Center, Miami, Florida, United States